CLINICAL TRIAL: NCT02503813
Title: Does Venous pCO2 Increase by 20 mmHg or More During Apnea Challenge Test?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Responsible Party: Principal Investigator, Alireza Fathi, MD, Director of Critical Care Transport, Assoicate Medical Director, PICU, MemorialCare Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 504-15
Record Dates: First submitted 2015-07-16; First posted 2015-07-21 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2015-07

CONDITIONS: Brain Death
Keywords: brain death; apnea challenge test
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Venous blood gas will be obtained at the same time points as arterial blood gas in the apnea challenge test.
  Interventions: Procedure: venous blood gas

INTERVENTIONS:
Procedure: venous blood gas — Venous blood gas will be measured at the time of arterial blood gas measurement.

SUMMARY:
One required examination for declaration of death by neurological criteria is the apnea challenge test. The apnea challenge test evaluates the medulla brainstem respiratory center response to a rise in CO2. The current guideline requires arterial sampling of CO2 and therefore either arterial puncture or arterial catheter placement for the examination. Arterial catheter is an invasive monitoring device and is not without complications. Recent studies have demonstrated that there is a direct correlation between peripheral venous and arterial blood gas measures and that peripheral venous CO2 measures may be used as alternatives to arterial CO2 measure.The purpose of this study is to evaluate brainstem response during the apnea challenge test to a rise in venous CO2 and correlate it with the rise in arterial measured CO2. The objective of this study is to demonstrate a similar rise between the venous and arterial CO2 during the apnea challenge test and eliminate the necessity of arterial blood sampling for the sole purpose of apnea challenge test in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 37 weeks gestation up to any adult age
2. Patients admitted to Pediatric Intensive Care unit (PICU), Neonatal Intensive Care Unit (NICU), Medical Intensive Care Unit (MICU) and Cardiothoracic Intensive Care Unit (CTICU)
3. Patients with irreversible brain injury where the attending physician will be performing death by neurological criteria examination as per hospital policy
4. Presence of arterial catheter or arterial blood sampling during apnea challenge test
5. Presence of central venous catheter or easily drawing peripheral intravenous catheter

Exclusion Criteria:

1. Age less or equal to 37 weeks gestation
2. Inability to perform apnea challenge test as determined by primary physician
3. Family request for Donation after Cardiac Death (DCD) or withdrawal of Life Sustaining Therapy
4. Bicarbonate infusion within 30 minutes of apnea challenge test

Min Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in venous blood CO2 during apnea challenge test | During apnea challenge test

SECONDARY OUTCOMES:
Change in End Tidal CO2 during apnea challenge test | During apnea challenge test

CONTACTS AND LOCATIONS:
Locations (1):
- Long Beach Memorial and Miller Children's & Women's Hospital Long Beach, Long Beach, California, United States

REFERENCES:
- [Result] Fathi A, Lake JL. Use of Venous Pco2 in Determination of Death by Neurological Criteria in Children. Pediatr Neurol. 2019 Apr;93:17-20. doi: 10.1016/j.pediatrneurol.2018.12.001. Epub 2018 Dec 19. PMID 30704867